CLINICAL TRIAL: NCT05432960
Title: International, Multi-Center, Double-blind, Randomized, Placebo-Controlled, Efficacy and Safety Clinical Study of RPH-104 in Adult Onset Still's Disease (AOSD)
Brief Title: Efficacy and Safety Clinical Study of RPH-104 in Adult Onset Still's Disease (AOSD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted according to the Sponsor's descision.
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Exacte Labs LLC (Industry); Ministry of Health, Russian Federation (Other Government); Scientific Center EFiS LLC (Unknown); Data Management 365 (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04018093
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Adult-Onset Still's Disease; AOSD
Keywords: RPH-104; subcutaneous
MeSH Terms: conditions — Still's Disease, Adult-Onset

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-104 (Experimental): The investigational product RPH-104 as SC injections at a dose of 160 mg on Day 0, Day 7, Day 21 and then once every 2 weeks (Q2W).
  Interventions: Biological: RPH-104
- Placebo (Placebo Comparator): placebo SC Q2W (equivalent to investigational product volume)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RPH-104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial
  Other Names: goflikicept; Arcerix
  Arms: RPH-104
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of RPH-104 when administered at a dose of 160 mg on Day 0, Day 7, Day 21 and then once every 2 weeks (Q2W) subcutaneous (SC) in patients with Adult Onset Still's Disease (AOSD). Furthermore, the study is scheduled to investigate pharmacokinetic (PK) and pharmacodynamic (PD) parameters of RPH-104.

DETAILED DESCRIPTION:
The overall study will include the following periods:

* screening period (up to 4 weeks) - the evaluation of patient compliance with inclusion/exclusion criteria.
* run-in period (29 weeks) - open-label administration of RPH-104 160 mg on Day 0, Day 7, Day 21 and then Q2W SC with gradual dose reduction with further complete withdrawal (if applicable) of the previous therapy with AOSD.

Baseline characteristics will be evaluated on Study Day 0. Assessment of efficacy (treatment response) and safety will be performed at Visit 2 (Day 7), Visit 3 (Day 21), Visit 4 (Day 35) and then every 4 weeks during the run-in period. A response to therapy during this period is the achievement of low activity/inactive disease including no exacerbations of AOSD.

The subjects who achieve and preserve low activity/inactive disease for at least 8 weeks under mono therapy with RPH-104 (i. e. previous therapy has been permanently discontinued) or combination of RPH-104 and GC at dose achieved in reduction (7.5 mg/day or less), stable for at least 4 weeks can be switched to the randomized withdrawal period.

• randomized withdrawal period (24 weeks) - blind SC administration of 160 mg of RPH-104 / equivalent volume of placebo Q2W depending on the distribution group in randomization; if the disease exacerbates during this period, a subject can be switched from placebo into a 53-week open-label therapy with RPH-104 (can be continued for 6 months in case of exacerbation as decided by the investigator).

Efficacy and safety assessment during the randomized withdrawal period will be performed every 4 weeks. During this period the investigational product/placebo will be administered to the subjects every 2 weeks - at visits to the study site - by the qualified medical staff (or a subject monitored by the staff) or at home by the subjects themselves. In case of self-administration of the investigational product/placebo by a subject during the randomized withdrawal period, additional conditions will be created to prevent from unblinding.

• safety follow-up period (8 weeks). The subjects who completed the randomized withdrawal period and the subjects who completed 53 weeks of resumed therapy (if applicable) and the subjects whose therapy was continued as decided by the investigator for 6 months after exacerbation in the randomized withdrawal period (for subjects from the investigational product group), or exacerbation during the resumed therapy - after the end of therapy will be switched into the safety follow-up period during which they will have to visit the study site for assessments in 2 and 8 weeks after the last dosing with the investigational products, thereafter their participation in the study will be considered completed.

The subjects who terminated therapy with RPH-104 early (for any reasons in any treatment period) will be prescribed with other products selected by the investigator and will have to make safety follow-up visits in 2 and 8 weeks after the last dosing with the investigational product.

Maximum possible duration of study per patient will be 144 weeks.

It is planned to randomize totally 36 patients with AOSD in the study (18 patients per group). Given potential withdrawal at the screening and during the run-in period, the number of screened patients (who signed informed consent) will be totally about 53 screened patients.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of voluntarily signed and dated Informed Consent Form to participate in this study.
2. Definite diagnosis of Still's disease made on the basis of Yamaguchi diagnostic criteria (Yamaguchi M., 1992).
3. A patient with AOSD (with inactive disease / low disease activity / exacerbation).
4. In case of current GCs administration, their doses should be stable for at least 2 weeks prior to Day 0. Maximum acceptable dose calculated as 1 mg/kg/day is up to 60 mg/day.
5. In case of on-going methotrexate (MTX) administration, the dose should be stable for at least 4 weeks prior to Day 0. Maximum acceptable dose is 30 mg/week. In case of withdrawal of previous MTX administration, it should be made at least 4 weeks before Day 0.
6. Ability and willingness of the subject, according to the reasonable investigator's judgment, to attend the study site at all scheduled visits, undergo the study procedures and follow the protocol requirements including subcutaneous injections by qualified site personnel.
7. Consent of female subjects with childbearing potential, defined as all females with physiological potential to conceive (except for those with absolute termination of menses to be determined retrospectively after 12 months of natural amenorrhea, i. e. amenorrhea with relevant clinical status, e. g. appropriate age) to use highly effective contraception throughout the study starting from the screening (signed Informed Consent Form) and for at least 8 weeks after discontinuation of the study product administration; and negative pregnancy test (serum test for chorionic gonadotropin).

OR Consent of male subjects leading active sexual life to use highly efficient contraceptive measures throughout the study starting from the moment of signing the Informed Consent Form and for at least 8 weeks after the study product discontinuation.

Highly effective contraceptive method is defined as follows:

* complete abstinence: if complies with patients' preferable and habitual way of life. Periodic abstinence (e. g. calendar, ovulation, symptothermal, post-ovulation methods) and interrupted intercourse are not acceptable contraception methods;
* surgical intervention for female sterilization: bilateral ovariectomy (with/without hysterectomy) or tubal ligation at least 6 weeks prior to the study therapy initiation. In case of ovariectomy only, the female reproductive status should be verified by further hormonal test;
* surgical intervention for male sterilization (with a relevant documented lack of the sperm in the post-vasectomy ejaculate) at least 6 months prior to screening. For female subjects, a vasectomized sexual partner should be the only partner;
* combination of any two of the following methods (a+b or a+c or b+c):

  1. oral, injection or implanted hormonal contraceptives; in case of oral contraceptives, the female subjects should administer the same product for at least 3 months prior to the study therapy;
  2. intrauterine device or contraceptive system;
  3. barrier contraception methods: a condom or occlusive cap (diaphragm or cervical cap/ vaginal fornix cap) with a spermicidal foam/ gel/ film/ cream/ vaginal suppository.

Exclusion Criteria:

1. Hypersensitivity to the investigational product (RPH-104) and/or its ingredients/excipients.
2. Previous administration of:

   * rilonacept - less than 6 weeks prior to Day 0 of the study;
   * canakinumab - less than 12 weeks prior to Day 0 of the study;
   * anakinra - less than 1 week prior to Day 0 of the study;
   * tumor necrosis factor alpha (TNF-a) antagonists, Interleukin 6 (IL-6) inhibitors - less than 12 weeks prior to Day 0 of the study;
   * Janus kinase inhibitors - less than 1 week prior to Day 0 of the study;
   * immunosuppressants (azathioprine, cyclosporin, mycophenolate mofetil, tacrolimus, sirolimus, mercaptopurine, etc., except for methotrexate) - less than 24 weeks prior to Study Day 0;
   * pulse therapy with GC (e. g., methylprednisolone 250-1000 mg/day intravenously or dexamethasone equivalent for 3 days) - less than 4 weeks (from the end of pulse therapy) to Study Day 0;
   * any other biological product - less than 5 half-lives prior to Study Day 0.
3. Administration of live (attenuated) vaccine less than 3 months prior to Visit 1 (study treatment period initiation) and/or necessity to use such vaccine within 3 months after the study therapy discontinuation. Live attenuated vaccines include viral vaccines against: measles, rubella, parotitis, varicella, rotavirus, influenza (as nasal spray), yellow fever, poliomyelitis (oral polio-vaccine), tuberculosis vaccine (BCG), typhoid (oral typhoid fever vaccine) and camp fever (epidemic typhoid vaccine). Immunocompetent family members should refuse to use oral polio-vaccine throughout the subject's participation in the study.
4. Conditions or signs which, according to the investigator, suggest impaired (reduced) immune response and/or significantly increase the risk of immunomodulating therapy including (but not limited to):

   * 4.1. active bacterial, fungal, viral or protozoal infection at screening onset;
   * 4.2. opportunistic infections and/or Kaposi's sarcoma at the screening period onset;
   * 4.3. chronic bacterial, fungal or viral infection requiring systemic therapy with parenteral products at the main screening period onset;
   * 4.4. human immunodeficiency viruses (HIV), hepatitis B or C.
5. Active infection of M. Tuberculosis, as per examination results: positive QuantiFERON-TB/SPOT.TB test at screening, chest X-ray findings confirming pulmonary tuberculosis during screening.

   * At discretion of certified tuberculosis specialist or pulmonologist specialized in diagnosing and treatment of tuberculosis, a patient with latent tuberculosis can be included in the study during the preventative treatment of latent tuberculosis infection with isoniazid or rifampicin (the choice of preventive therapy is made by a phthisiatrician, taking into account contraindications, drug interactions and risks of adverse reactions in a particular patient).
6. Any other relevant concomitant diseases (cardiovascular, nervous, endocrine, urinary, gastrointestinal, hepatic disorders, hemostatic disorders, other autoimmune diseases, etc.) or conditions which, according to the investigator's judgment, may affect the subject's participation or well-being in the study and/or distort assessment of the study results.
7. History of organ transplantation or necessity in transplantation at the screening onset.
8. Any malignancies during the screening period or for 5 years before screening except for non-metastatic basal cell and squamous cell skin cancer after total resection or in situ carcinoma of any type after total resection.
9. Psychiatric disorders which, according to the justified investigator's judgment, may affect the subject participation in the study and his/her ability to follow the protocol procedures.
10. Pregnancy or breast-feeding.
11. History of alcohol or psychoactive substances abuse, according to the investigator's evaluation.
12. Severe renal failure: Cockroft-Gault creatinine clearance (ClCr) < 30 mL/min.
13. Any of the deviations in the laboratory tests below:

    * absolute neutrophil count < 1.5 х 10^9/L;
    * white blood cells (WBC) count < 3.5 х 10^9/L;
    * platelet count < 100 х 10^9/L;
    * hemoglobin level ≤ 80 g/L;
    * glycated hemoglobin (HbA1c) ≥ 8 %);
    * alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 8.0 x upper limits of normal (ULN);
    * AST and/or AST > 3 x ULN with increased bilirubin > 1.5 x ULN;
    * bilirubin > 1.5 x ULN (except for confirmed Gilbert's disease).
14. Uncontrolled diabetes mellitus.
15. Concomitant participation in other clinical studies at the screening onset or administration of any unauthorized (investigational) products less than 4 weeks or 5 half-life periods (whichever is longer) before Visit 1 (treatment initiation in the study).
16. Macrophage activation syndrome (MAS) in the history or suspected at screening.
17. MAS diagnosed within the last 2 months prior to Day 0.
18. Previous participation in this clinical study if at least one dose of the investigational product has been received.

    * MAS criteria: Fever and hyperferritinemia > 684 ng/mL combined with at least 2/4 criteria:

      * Decreased platelet count ≤181 х 10^9/L
      * Elevated AST level > 48 U/L
      * Triglyceride elevation >156 mg/dL
      * Decreased fibrinogen ≤ 360 mg/dL Laboratory abnormalities should not be related with other comorbid conditions of the patient, such as immune-mediated thrombocytopenia, infectious hepatitis, visceral leishmaniasis, or familial hyperlipidemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Time (number of days) to exacerbation during 24 weeks after randomization while taking RPH-104 vs placebo in patients with AOSD | from randomization (visit 16, week 29) to exacerbation, up to week 53
  The criteria for exacerbation are (more than 2 criteria or worsening of more than 2 previous criteria):
  * fever (body temperature ≥ 38.0 °C) due to AOSD during a week before the visit;
  * rash typical of AOSD;
  * clinical disease activity index (CDAI) > 2.8 for subjects with inactive disease; > 10 for subjects with low disease activity*;
  * sore throat*;
  * pericardial effusion ≥ 7 mm*;
  * pleuritis*;
  * chest pain > 3 numeric rating scale (NRS)*;
  * C-reactive protein (CRP) > 5 mg/L*;
  * aminotransferase (ALT, AST) level > 3 x upper limits of normal (ULN)*;
  * leukocyte count > 10 x 10^9/L with > 80 % polymorphonuclear neutrophils*;
  * ferritin level > 3 x ULN*;
  * Patient's Global Assessment (PtGA) worsening by 2 cm and more;
  * Physician's Global Assessment (PGA) worsening by 2 cm and more;
  * myalgia*;
  * hepatomegaly*;
  * splenomegaly*;
  * lymphadenopathy*. * Increase/presence of noted signs due to other reason than AOSD should not be considered in the activity assessment for AOSD exacerbation.

SECONDARY OUTCOMES:
Proportion of patients from RPH-104 group who developed AOSD exacerbation during 24 weeks after randomization vs placebo | up to week 53
  The criteria for exacerbation are (more than two criteria or worsening of more than two previous criteria):
  * fever, i. e. body temperature ≥ 38.0 °C due to AOSD lasting at least two consecutive days;
  * rash typical of AOSD;
  * sore throat*;
  * pericardial effusion ≥ 7 mm*;
  * pleuritis*;
  * aminotransferase (ALT, AST) level > 3 x ULN*;
  * leukocyte count > 15 x 10^9/L*;
  * ferritin level > 3 x ULN*;
  * myalgia*;
  * hepatomegaly*;
  * splenomegaly*;
  * lymphadenopathy*;
  * pneumonia*;
  * arthritis*. * Increase/presence of noted signs due to other reason than AOSD should not be considered in the activity assessment for AOSD exacerbation.
Proportion of patients who developed AOSD exacerbation during the run-in period | up to week 29
  The criteria for exacerbation are (more than two criteria or worsening of more than two previous criteria):
  * fever, i. e. body temperature ≥ 38.0 °C due to AOSD lasting at least two consecutive days;
  * rash typical of AOSD;
  * sore throat*;
  * pericardial effusion ≥ 7 mm*;
  * pleuritis*;
  * aminotransferase (ALT, AST) level > 3 x ULN*;
  * leukocyte count > 15 x 10^9/L*;
  * ferritin level > 3 x ULN*;
  * myalgia*;
  * hepatomegaly*;
  * splenomegaly*;
  * lymphadenopathy*;
  * pneumonia*;
  * arthritis*. * Increase/presence of noted signs due to other reason than AOSD should not be considered in the activity assessment for AOSD exacerbation.
Proportion of patients with fever resolution | up to Day 14
  Proportion of patients with fever resolution during the run-in treatment period.
  Fever resolution means body temperature < 38.0 °C
Proportion of patients with Simple disease activity index (SDAI) ≤ 3.3 | up to Day 203
  Proportion of patients with SDAI ≤ 3.3 during the run-in treatment period.
  SDAI is the sum of five parameters:
  * Physician's Global Assessment (PGA) and
  * Patient's Global Assessment (PtGA)
  * C-Reactive Protein (CRP) level*
  * Number of joints with active arthritis (based on an assessment of 28 joints): Tender Joint Count (TJC) (0-28) + Swollen Joint Count (SJC) (0-28) + PtGA (Visual analogue scale (VAS) in cm) + PGA (VAS) + CRP (mg/dl) The maximum score is 86 with high disease activity (the worst outcome). *Another cause for the elevated CRP must be ruled out.
Proportion of patients with CDAI 3.3 - 11 | up to Day 203
  Proportion of patients with CDAI 3.3 - 11 during the run-in treatment period.
  CDAI will be calculated using the following formula: CDAI = tender joint number (TJN) (0-28) + swollen joint number (SJN) (0-28) + Patient Global Assessment of Disease Activity (Visual analogue scale (VAS) in cm) + Physician Global Assessment (VAS in cm).
  CDAI Range: 0 - 76, with a decrease from baseline indicating improvement.
Proportion of patients with a decrease in modified Pouchot score (mPouchot) score of at least 3 points or a decrease in mPouchot score of at least 1 point, provided that mPouchot score ≤4 at baseline (Day 0), during the run-in treatment period | up to Day 203
  mPouchot score is calculated by assigning 1 point to each of these items:
  * fever (body temperature ≥ 38.0 °C due to AOSD);
  * rash typical of AOSD (according to data of physical examination);
  * number of joints with active arthritis (0 to 68/66 joints)*;
  * sore throat (according to complaints as of examination)*;
  * pericardial effusion (Echocardiography)*;
  * pleuritis (ultrasound examination of the lungs)*;
  * aminotransferase (ALT, AST) activity*;
  * leukocyte count*;
  * ferritin level*;
  * myalgia (according to complaints as of examination)*;
  * hepatomegaly (ultrasound examination of the abdominal organs)*;
  * lymphadenopathy (physical examination)*;
  * Pneumonia (chest X-ray data)*. The maximum score is 12 points with high disease activity (the worst outcome). Hepatomegaly and aminotransferase levels are 1 point.
    * For noted signs, which are not AOSD-specific, other reason for their increase/presence should be considered in the activity assessment for AOSD exacerbation.
Proportion of patients with clinically significant reduction in joint manifestations | up to Day 203
  Proportion of patients with clinically significant reduction in joint manifestations - SDAI reduced by at least 7 points from baseline (Day 0), during the run-in treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (4):
- Russia (4):
  - Research Institute of Rheumatology. V.A. Nasonova, Moscow
  - Clinic of Nephrology, Internal and Occupational Diseases. EAT. Tareeva, University Clinical Hospital No. 3, Moscow
  - State Budgetary Institution of Healthcare Leningrad Regional Clinical Hospital, Department of Rheumatology, Saint Petersburg
  - FGBU "National Medical Research Center named after V.A. Almazov", Ministry of Health of the Russian Federation, Department of Rheumatology, Saint Petersburg